CLINICAL TRIAL: NCT03078036
Title: BREAKOUT -International Breast Cancer Biomarker, Standard of Care and Real World Outcomes Study
Brief Title: International Breast Cancer Biomarker,Standard of Care and Real World Outcomes Study
Acronym: BREAKOUT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles; University of Tubingen - Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: D0816R00012
Record Dates: First submitted 2017-02-10; First posted 2017-03-13 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: HER2-ve metastatic breast cancer; gBRCA, sBRCA and HRR gene mutations
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole Blood and Archived Tumor Specimen (e.g. tumor tissue)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Human epidermal growth factor receptor 2 negative metastic breast cancer patients who have started 1st line systemic cytotoxic chemotheraphy and are considered to have exhausted hormone therapy options (if HR+ve), per investigator's opinion.
  Interventions: Genetic: Germline BRCA Test (blood); Genetic: FoundationOne Dx Genomic Profile (archival Tumour Specimen); Other: Follow-up

INTERVENTIONS:
Genetic: Germline BRCA Test (blood) — If unavailable from the patient medical records, gBRCA gene mutation status will be tested as aligned to local clinical practice using a blood sample obtained preferably during routine clinical practice. (Note: Blood samples may be shipped to a central laboratory for testing and storage, based on local regulations for shipment of blood samples.)
Genetic: FoundationOne Dx Genomic Profile (archival Tumour Specimen) — Archival tumour specimen will be requested from all patients in the informed consent, but is not required for study enrolment (optional consent). Where sufficient archival tumour specimen is available and patients have consented to tumour specimen testing, FoundationOne Dx genomic profiling may take place as follows:
  * Tumour Specimen: Acceptable samples include formalin-fixed, paraffin embedded (FFPE) tissue (preferred) or FFPE specimens, including core needle biopsies, fine-needle aspirates and effusion cytologies.
  * Tumour Testing (optional): archival tumour specimens, where available, will be tested for mutations in HRR genes including BRCA1 and BRCA2 and other genomic alterations using the FoundationOne Dx genomic profile.
Other: Follow-up — Patients who test positive for a gBRCA gene mutation, and/or sBRCA or other HRR gene mutations (optional testing), will be followed prospectively for assessment of treatment patterns and associated clinical outcomes up to 30-months.
  - Patients who test negative for gBRCA gene mutations, sBRCA and other HRR gene mutations, no further data will be collected post baseline. Patients presenting other genomic alterations that are identified by the FoundationOne Dx genomic profile will not continue beyond baseline as part of this study.

SUMMARY:
BREAKOUT -International Breast Cancer Biomarker, Standard of Care and Real World Outcomes Study BREAKOUT is a prospective cross-sectional cohort study of human epidermal growth factor receptor 2 negative metastatic breast cancer patients who have started 1st line systemic cytotoxic chemotherapy. The study will estimate the prevalence of germline breast cancer susceptibility gene in an otherwise unselected population, describe the treatments administered and estimate the associated clinical outcomes of overall survival and progression-free survival amongst mutation carriers within the context of a low poly ADP ribose polymerase inhibitor treatment setting. Other exploratory analyses may be undertaken to describe somatic breast cancer susceptibility gene and other homologous recombination repair gene mutations.

DETAILED DESCRIPTION:
Background/Rationale: Within the setting of metastatic human epidermal growth factor receptor 2 negative (HER2-ve) breast cancer limited epidemiological data exist on the prevalence of pathogenic mutations of breast cancer susceptibility gene (BRCA) and other homologous recombination repair (HRR) genes. There are also limited data on the treatments and clinical outcomes of patients with such germline and somatic genetic profiles, particularly within this setting. This epidemiologic study will estimate the prevalence of germline breast susceptibility gene (gBRCA) mutations among metastatic HER2-ve patients who have commenced 1st line systemic cytotoxic chemotherapy and, at that time, are considered to have exhausted hormone therapy options (if hormone receptor positive [HR+ve]), per investigator's opinion. Among those patients with a gBRCA gene mutation, treatment patterns and clinical outcomes will be described. This study may also explore the prevalence of somatic BRCA (sBRCA) mutations and other HRR gene mutations among metastatic HER2-ve patients who have commenced 1st line systemic cytotoxic chemotherapy. The treatment patterns and clinical outcomes may be described among those patients with a sBRCA gene mutation and those with other HRR gene mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed, written and dated informed consent.
2. Adult females (according to the age of majority/adulthood as defined by local regulations).
3. Histologically or cytologically confirmed HER2-ve breast cancer with evidence of metastatic disease.
4. Initiated treatment with 1st line systemic cytotoxic chemotherapy (not hormonal therapy) for metastatic breast cancer in the last 90 days and, at that time, are considered to have exhausted hormone therapy options (if HR+ve).

Exclusion Criteria:

1. Previous enrolment in this study.
2. Involvement in the planning and/or conduct of this study (applies to both AstraZeneca staff and/or staff at the study site).
3. Current participation in a clinical study with an investigational oncology product.
4. Previous PARPi therapy, including, but not limited to, participation in a previous clinical study that included PARPi therapy.
5. Current commencement of PARPi treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Centers for primary care of metastatic HER2-ve breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 873 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
BRCA Mutational status (BRCA1 mutated and/or BRCA2 mutated or BRCA wild type). | At one time point at inclusion in the study up to 12 months after the beginning of the study.
  The prevalence of gBRCA gene mutations will be evaluated by calculating the proportion of patients that test positive for a gBRCA gene mutation (BRCA1 mutated and/or BRCA2 mutated).

SECONDARY OUTCOMES:
Descriptive statistics for treatments administered by line of therapy from 1st line metastatic breast cancer. | 2.5 years (30 months) since the beginning of the study.
  Treatment patterns will be described by line of therapy. Treatment combinations, number of cycles per line, schedules, durations, and reason for discontinuation will be summarized descriptively.
Progression free survival by line of therapy | 2.5 years (30 months) since the beginning of the study.
  Progression free survival (in months) for each line of treatment, defined as the time from the date of start of each line of treatment to the documented date of progression as determined by the investigator (radiologic or symptomatic), or death from any cause in the absence of progression.
Overall survival by line of therapy | 2.5 years (30 months) since the beginning of the study.
  Overall survival (OS) defined as the time from the start date of first line chemotherapy in the metastatic setting until the date of death due to any cause, assessed up to 30 months. In addition, OS since diagnosis of metastatic breast cancer and OS since the start of each subsequent therapy will be estimated.

CONTACTS AND LOCATIONS:
Locations (97):
- United States (13):
  - Research Site, Santa Barbara, California
  - Research Site, Denver, Colorado
  - Research Site, Hialeah, Florida
  - Research Site, Dallas, Texas
  - Research Site, Denton, Texas
  - Research Site, Flower Mound, Texas
  - Research Site, Houston, Texas
  - Research Site, Paris, Texas
  - Research Site, San Antonio, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Newport News, Virginia
  - Research Site, Vancouver, Washington
  - Research Site, Wenatchee, Washington
- Australia (3):
  - Research Site, Redcliffe, Queensland
  - Research Site, Kurralta Park, South Australia
  - Research Site, Ballarat, Victoria
- Bulgaria (3):
  - Research Site, Dobrich
  - Research Site, Rousse
  - Research Site, Sofia
- Canada (4):
  - Research Site, Kingston, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Québec
- Research Site, Tübingen, Germany
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Szolnok
- Italy (5):
  - Research Site, Carpi, Modena
  - Research Site, Castellanza, Varese
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Reggio Emilia
- Japan (7):
  - Research Site, Kamogawa-shi, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Sendai, Miyagi
  - Research Site, Osaka, Osaka
  - Research Site, Chūōku, Tokyo-To
- Poland (7):
  - Research Site, Brzozów
  - Research Site, Opole
  - Research Site, Warsaw
  - Research Site, Wałbrzych
  - Research Site, Wieliszew
  - Research Site, Wroclaw
  - Research Site, Żory
- Russia (7):
  - Research Site, Chelyabinsk
  - Research Site, Krasnodar
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Tomsk
- South Korea (5):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Seoul
  - Research Site, Ulsan
- Spain (8):
  - Research Site, Terrassa, Barcelona
  - Research Site, A Coruña, La Coruña
  - Research Site, Alcorcón, Madrid
  - Research Site, San Sebastián de los Reyes, Madrid
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Girona
  - Research Site, Huelva
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (12):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Diyarbakır
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Sakarya
  - Research Site, Samsun
  - Research Site, Tekirdağ
  - Research Site, Trabzon
  - Research Site, Van
- United Kingdom (13):
  - Research Site, Huntingdon, Cambridgeshire
  - Research Site, Peterborough, Cambridgeshire
  - Research Site, Truro, Cornwall
  - Research Site, Derby, Derbyshire
  - Research Site, Exeter, Devon
  - Research Site, Worthing, East Sussex
  - Research Site, London, Greater London
  - Research Site, Blackpool, Lancashire
  - Research Site, Lancaster, Lancashire
  - Research Site, Stoke-on-Trent, Staffordshire
  - Research Site, Warwick, Warwickshire
  - Research Site, Wolverhampton, West Midlands
  - Research Site, Huddersfield, West Yorkshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koh SJ, Ohsumi S, Takahashi M, Fukuma E, Jung KH, Ishida T, Dai MS, Chang CH, Dalvi T, Walker G, Bennett J, O'Shaughnessy J, Balmana J. Prevalence of mutations in BRCA and homologous recombination repair genes and real-world standard of care of Asian patients with HER2-negative metastatic breast cancer starting first-line systemic cytotoxic chemotherapy: subgroup analysis of the global BREAKOUT study. Breast Cancer. 2022 Jan;29(1):92-102. doi: 10.1007/s12282-021-01283-4. Epub 2021 Aug 31. PMID 34467476
- [Derived] O'Shaughnessy J, Brezden-Masley C, Cazzaniga M, Dalvi T, Walker G, Bennett J, Ohsumi S. Prevalence of germline BRCA mutations in HER2-negative metastatic breast cancer: global results from the real-world, observational BREAKOUT study. Breast Cancer Res. 2020 Oct 27;22(1):114. doi: 10.1186/s13058-020-01349-9. PMID 33109210
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816R00012&attachmentIdentifier=fb200c6c-0fb4-423a-aedc-f0b69c5717fc&fileName=D0816R00012_Study_Report_Synopsis_FINAL_Redacted.pdf&versionIdentifier=